CLINICAL TRIAL: NCT02260375
Title: THIRD-PARTY BONE MARROW-DERIVED MESENCHYMAL STROMAL CELLS TO INDUCE TOLERANCE IN LIVER TRANSPLANT RECIPIENTS
Brief Title: MSC Therapy in Liver Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Monia Lorini (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor-Investigator, Monia Lorini, EC Secretary, A.O. Ospedale Papa Giovanni XXIII
Organization: A.O. Ospedale Papa Giovanni XXIII (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC liver transplant tolerance; 2014-001531-37 (EudraCT Number)
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Liver Transplant Rejection
Keywords: Mesenchymal stromal cells; liver transplantation; tolerance.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesenchymal Stromal Cells (MSC) (Experimental): A single intravenous infusion (1-2 millions of MSCs per kilogram body weight) of ex-vivo expanded third-party MSC (from healthy donors) will be performed in patients assigned to the MSC procedure in addition to the liver transplantation.
  Interventions: Biological: Mesenchymal Stromal Cells
- No treatment. (No Intervention)

INTERVENTIONS:
Biological: Mesenchymal Stromal Cells
  Arms: Mesenchymal Stromal Cells (MSC)

SUMMARY:
The general aim of the present study is to test a cell therapy with third-party allogeneic ex-vivo expanded MSCs as a strategy to induce tolerance in liver transplant recipients. MSCs will be prepared accordingly to established protocols , starting from diagnostic samples of bone marrow aspirates (2-5 mL) or using the remnants in the bag and filter at the end of the bone marrow infusions. From these samples, MSCs will be expanded in GMP approved facilities and used for the present study in patients undergoing liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

For this study, the following inclusion criteria should be fulfilled before starting withdrawal of drugs after 1 year post-transplant:

* First liver transplant
* Capable of understanding the purpose and risk of the study
* Written informed consent

Exclusion Criteria:

* Specific contraindication to MSC infusion
* Any clinical relevant condition that might affect study participation and/or study results
* Pregnant women and nursing mothers
* Unwillingness or inability to follow the study protocol in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | Changes from baseline up to 120 month.
  At each visit overall clinical condition of the patient will be evaluated and any adverse event will be recorded.
Liver tissue mRNA level of Transferrin receptor CD71 (TFRC) and Hepcidin antimicrobial peptide (HAMP) genes | At 12 and 60 month.
Circulating naive and memory T cell conts (CD45RA/CD45RO)(flow cytometry analysis) | Changes from baseline at 6 and 12 months after transplant, then every 6 months till the first 3 years after transplant and then yearly up to 120 month.
T-cell function in mixed lymphocyte reaction | Changes from baseline at 6 and 12 months after transplant, then every 6 months till the first 3 years after transplant and then yearly up to 120 month.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Chair — A.O. Ospedale Papa Giovanni XXIII; Norberto Perico, MD, Study Director — IRCCS-Istituto di Ricerche Farmacologiche M. Negri; Michele Colledan, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII; Stefano Fagiuoli, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII; Martino Introna, MD, Principal Investigator — Laboratorio G.Lanzani, Bergamo, Italy; Alessandro Rambaldi, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII; Antonio Pinna, MD, Principal Investigator — Policlinico S. Orsola Bologna, Italy; Claudio Velati, MD, Principal Investigator — Policlinico S. Orsola Bologna, Italy
Locations (6):
- Italy (6):
  - U.S.C Nefrologia e Dialisi, Bergamo
  - USC Chirurgia Generale III, Bergamo
  - USC Ematologia, Bergamo
  - USC Gastroenterologia, Bergamo
  - Servizio di Immunoematologia e Medicina Trasfusionale, Bologna
  - Unità Chirurgia Generale e Trapianti, Bologna

REFERENCES:
- [Derived] Casiraghi F, Perico N, Podesta MA, Todeschini M, Zambelli M, Colledan M, Camagni S, Fagiuoli S, Pinna AD, Cescon M, Bertuzzo V, Maroni L, Introna M, Capelli C, Golay JT, Buzzi M, Mister M, Ordonez PYR, Breno M, Mele C, Villa A, Remuzzi G; MSC-LIVER Study Group. Third-party bone marrow-derived mesenchymal stromal cell infusion before liver transplantation: A randomized controlled trial. Am J Transplant. 2021 Aug;21(8):2795-2809. doi: 10.1111/ajt.16468. Epub 2021 Feb 22. PMID 33370477